CLINICAL TRIAL: NCT01364844
Title: A Phase 1, Open-Label, Multiple-Escalating-Dose Study of DS-7423, an Orally Administered Dual PI3K/mTOR Inhibitor, in Subjects With Advanced Solid Tumors
Brief Title: Safety and Tolerability of DS-7423 in Subjects With Advanced Solid Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS7423-A-U101
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Solid Tumor; Colorectal Cancer; Endometrial Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Endometrial Neoplasms | interventions — DS7423

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DS7423 (Experimental)
  Interventions: Drug: DS-7423

INTERVENTIONS:
Drug: DS-7423 — oral capsule 1mg, 8mg, 48mg, and 80mg strengths administered once daily

SUMMARY:
This will be a Phase 1, open-label study of DS-7423 to assess its safety and tolerability, identify a RP2D, (recommended Phase 2 Dose) and assess its Pharmacokinetics (PK) (what your body does to process the drugs and how your body gets them out of your system.) and pharmacodynamics (PDy) (Pharmacodynamics is a study of what a drug does to your body) properties in subjects with advanced solid malignant tumors. This study will include 2 parts: part 1-Dose Escalation and part 2-Dose Expansion.

Study Hypothesis: DS-7423 will be safe and tolerable, and will exhibit acceptable PK and PDy properties in subjects with advanced solid malignant tumors for whom standard therapy has failed or for whom no standard therapy exists.

DETAILED DESCRIPTION:
Part 1 : Dose-escalation of DS-7423 to determine maximum tolerated dose (MTD) in subjects with advanced solid tumors Part 2 : Dose Expansion: The purpose of Part 2 of this clinical research study is to confirm the safety and tolerability of the MTD of DS-7423 identified in Part 1, and measure the effects of DS-7423 on your cancer. Part 2 will be conducted in subjects with advanced colorectal or endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* A pathologically documented advanced solid malignant tumor refractory to standard treatment or for which no standard treatment is available
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Have adequate bone marrow function, defined as:

Platelet count >= 100 X 10^9/L Hemoglobin (Hb) level >= 9.0 g/dL ANC >= 1.5 X 10^9/L - Have adequate renal function, defined as: Creatinine clearance >= 60 mL/min, as calculated using the modified Cockroft Gault equation, ([{140 - age in yrs} x {actual weight in kg}] divided by [{72 x serum creatinine in mg/dL} multiply by 0.85 if female]), or creatinine =< 1.5 X ULN

- Have adequate hepatic function, defined as: AST/ALT levels =< 3 X ULN (if liver metastases are present, =< 5 X ULN) Bilirubin =< 1.5 X ULN

- Have adequate blood clotting function, defined as: Prothrombin time and activated partial thromboplastin time =< 1.5 X ULN

* Subjects should be able to provide written informed consent, comply with protocol visits and procedures, be able to take oral medication, and not have any active infection or chronic comorbidity that would interfere with therapy
* Subjects (male and female) of childbearing potential must agree to use double-barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug
* Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an Institutional Review Board (IRB) approved informed consent form (ICF) (including Health Insurance Portability and Accountability Act (HIPAA) authorization, if applicable) before performance of any study-specific procedures or tests
* Subjects must be willing to provide available preexisting diagnostic or resected tumor samples, such as formalin-fixed paraffin-embedded sections. Providing fresh tumor biopsy is optional for subjects in dose escalation cohorts. Pre- and posttreatment biopsies are optional for all the subjects in Dose Escalation cohorts but required for those in Dose Expansion cohorts

Additional Inclusion Criteria for Part 2 (Dose Expansion)

* A pathologically documented advanced colorectal or endometrial cancer, with measurable disease based on RECIST criteria, Version 1.1, that is refractory to standard treatment
* Agree to undergo pre- and posttreatment tumor biopsies

Exclusion Criteria:

* History of second malignancy and primary central nervous system malignancies, except adequately treated nonmelanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated, with no evidence of disease for >= 3 years
* Gastrointestinal diseases that could affect the absorption of DS-7423
* Subjects with a fasting glucose > 126 mg/dL (> 7 mmol/L)
* History of diabetes mellitus (Type I or II) or hemoglobin A1c (HbA1c) > 7.0%
* Tested positive for hepatitis B or C serological markers (HBsAg or antiHCV)
* Recipient of live vaccine within 1 month of or during study drug treatment
* Concomitant use of chronic systemic corticosteroids
* Subjects requiring daily supplemental oxygen
* Recipient of a stem cell or bone marrow transplant
* Has a concomitant medical condition that would increase the risk of toxicity, in the opinion of the investigator or sponsor
* Clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 4 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment (2 weeks for stereotactic radiotherapy)
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI CTCAE, Version 4.0, grade =< 1 or baseline. Subjects with chronic grade 2 toxicities may be eligible per the discretion of the investigator or sponsor (eg, grade 2 chemotherapy-induced neuropathy)
* Systemic treatment with anticancer therapy, antibody-based therapy, retinoid therapy, or hormonal therapy within 3 weeks before study drug treatment; or treatment with nitrosoureas or mitomycin C within 6 weeks before study drug treatment; or treatment with small-molecule targeted agents within 2 weeks, or 5 half-lives before study drug treatment, whichever is longer. Previous and concurrent use of hormone replacement therapy, the use of gonadotropin-releasing hormone modulators for prostate cancer, and the use of somatostatin analogs for neuroendocrine tumors are permitted if such therapy has not been changed within 60 days before study drug treatment
* Therapeutic radiation therapy or major surgery within 4 weeks before study drug treatment or palliative radiation therapy within 2 weeks before study drug treatment
* Participation in a clinical study within 3 weeks (2 weeks or 5 half-lives, whichever is longer, for small-molecule targeted agents) before study drug treatment, or current participation in other investigational procedures
* Concomitant treatment with strong inducers or strong inhibitors of cytochrome P450 (CYP) 3A4/5, and CYP2C8
* Prolongation of corrected QT interval by Fridericia's method (QTcF) at rest, where the mean QTcF interval is > 450 millisecond (ms) for males and > 470 ms for females based on triplicate ECG
* Pregnant or breastfeeding
* Substance abuse or medical, psychological, or social conditions that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results
* Prior NCI CTCAE, Version 4.0, grade 3/4 toxicity from a dual phosphatidylinositol 3 kinase (PI3K)/mammalian target of rapamycin (mTOR) inhibitor (including, but not limited to, BEZ-235, XL765, GDC-0980, SF1126, GSK2126458, PF4691502, and PF05212384), requiring dose reduction and/or study discontinuation

Additional Exclusion Criteria for Part 2 (Dose Expansion)

- Prior treatment with a dual PI3K/ mTOR inhibitor (including, but not limited to, BEZ-235, XL765, GDC-0980, SF1126, GSK2126458, PF4691502, and PF05212384)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 30 days after last dose
  All adverse events will be graded according to the NCI-CTCAE, version 4.0

SECONDARY OUTCOMES:
Plasma pharmacokinetics of DS-7423 | Cycle 1 - days 1, 2, 8, and 15; Cycle 2 - day 1; end of study
  The various pharmacokinetic parameters will be calculated from plasma concentrations of DS-7423 using non-compartmental analyses.
Effects of DS-7423 on glucose metabolism | Cycle 1 Days 1, 2, and 15; and end-of-study
  The effects of DS-7423 on glucose metabolism will be determined by measuring glucose and C-peptide levels
Pharmacodynamic effects of DS-7423 in surrogate tissues | Cycle 1 Days 1, 2, and 15
  The pharmacodynamic effects of DS-7423 will be determined by measuring phosphorylation of Akt in platelet-rich plasma
Pharmacodynamic effects of DS-7423 in tumors | Baseline and Cycle 1 Day 4
  The pharmacodynamic effects of DS-7423 will be determined by measuring tumor glucose uptake using (18F) fluorodeoxyglucose-positron emission tomography
Part 2 - Objective response rate in subjects with advanced colorectal and endometrial cancer | Baseline and every 2 cycles of treatment for the first 8 cycles and then every 3 cycles thereafter until study drug discontinuation
  Objective response rate = the sum of complete response [CR] and partial response [PR] rates as measured using Response Evaluation Criteria in Solid Tumors (RECIST) criteria Version 1.1
Part 2 - Pharmacodynamic effects of DS-7423 in tumors | Baseline and Cycle 1 Day 15
  The pharmacodynamic effects of DS-7423 in tumors will be determined by measuring Akt, ribosomal protein S6 (S6), and proline-rich Akt substrate, 40 kDA (PRAS40) phosphorylation in pre- and posttreatment tumor biopsies

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee